CLINICAL TRIAL: NCT04806113
Title: COVID-19 Vaccine in Immunosuppressed Adults With Autoimmune Diseases
Acronym: COVIAAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: CHU de Quebec-Universite Laval (Other); Ministere de la Sante et des Services Sociaux (Other)
Responsible Party: Principal Investigator, Ines Colmegna, MD, Associate Professor, Rheumatology - Department of Medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MP-37-2021-7562
Record Dates: First submitted 2021-03-12; First posted 2021-03-19 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Covid19; Rheumatic Diseases; Rheumatoid Arthritis; SLE
MeSH Terms: conditions — COVID-19; Rheumatic Diseases; Arthritis, Rheumatoid | interventions — 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Intervention Model Description: Non-randomized, open label, comparative clinical trial with pragmatic features.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vaccine (Other): Study participants (People with rheumatic diseases and age matched controls).
  Interventions: Biological: Moderna COVID-19 vaccine

INTERVENTIONS:
Biological: Moderna COVID-19 vaccine — Two doses from the Moderna vaccine will be administered intramuscularly. The time between dose 1 and dose 2 of the vaccine will be 28 days.

SUMMARY:
This study will evaluate the Moderna RNA-based COVID-19 vaccine currently approved by Health Canada in people with rheumatic diseases. This study will help understand what the side effects of the vaccine in these patients are, and what is their capacity to develop antibodies that may confer protection from the COVID-19 disease.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, local reactions (reactogenicity), capacity to form antibodies against the coronavirus (immunogenicity) and long-term persistence of those antibodies following two doses of a Health Canada approved RNA-based COVID-19 vaccine in patients with rheumatic diseases.

Two doses from the Moderna vaccine will be administered intramuscularly. The time between dose 1 and dose 2 of the vaccine will be 28 days.

This research study will recruit 220 participants (165 patients and 55 healthy controls), men and women, aged 18 years or older.

ELIGIBILITY:
Inclusion Criteria (all of the following):

1. Adults ages 18 years and older;
2. For the cases, established diagnosis of:

   1. RA done by a rheumatologist according to the 2010 American College of Rheumatology (ACR) /European League Against Rheumatism (EULAR) criteria, OR
   2. SLE done by a rheumatologist according to the 1997 revised ACR criteria and/or the 2013 SLICC lupus classification criteria and/or the 2019 EULAR/ACR criteria;
3. For the cases, stable treatment (≥3 months prior to enrollment for biologics/small molecules and MMF; >3 weeks of a specific dose in case of steroids);
4. For the controls, people without a diagnosis of a chronic rheumatic disease who can have comorbidities as in patients with rheumatic diseases;
5. Able to comprehend the investigational nature of the protocol and provide informed consent;
6. Male or non-pregnant female;
7. Women of childbearing potential must agree to use at least one acceptable primary form of contraception.

Exclusion Criteria (any of the following):

1. Positive pregnancy test either at screening or just prior to each vaccine administration.
2. Any medical disease or condition that, in the opinion of the site Principal Investigator (PI) or appropriate sub-investigator, precludes study participation.
3. Acute illness, as determined by the site PI or appropriate sub-investigator, with or without fever [oral temperature >38.0°C (100.40F)] within 72 hours prior to each vaccination.
4. Diagnosis of hepatitis B, hepatitis C virus, or human immunodeficiency virus (HIV).
5. History of hypersensitivity or severe allergic reaction (e.g., anaphylaxis, generalized urticaria, angioedema, other significant reaction) to any previous licensed or unlicensed vaccines.
6. Participation in another clinical trial or plan to do so during the study. If a patient was on a drug trial, recruitment could occur following 2 half-lives of the study drug.
7. Vaccines within the 2 weeks prior to any dose of COVID-19 vaccine or until 30 days after any dose of COVID-19 vaccine.
8. Lactating female.
9. Immunoglobulin therapy or blood products within the past month.
10. Prior diagnosis of COVID-19 in the past 3 months.
11. Planned changes in baseline drug treatments (except prednisone) for rheumatic diseases prior to D57.
12. For patients required to be on cohort 8: Planned reduction of prednisone dose below 10 mg prior to D21.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2021-06-13 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Frequency and grade of each solicited local and systemic adverse events (AEs) | during a 7-day follow-up period post each vaccination
Frequency and grade of any unsolicited AEs (including 'significant disease flares'*) | during the 28-day follow-up period post-each vaccine dose.
  * 'Significant' disease flares: defined as worsening of clinical disease activity documented by the treating physician and requiring intensification of therapy.

SECONDARY OUTCOMES:
Geometric mean titer (GMT) of antibody | at Day 57
Percentage of patients who seroconverted | baseline and Day 57
  defined as a 4-fold increase in antibody titer
Geometric mean fold rise (GMFR) in IgG titer | baseline and Day 57

OTHER OUTCOMES:
Geometric mean titer (GMT) of antibody | Day 28
  post-first vaccine dose
Geometric mean titer (GMT) of neutralizing antibody | Day 57
CD4 and CD8 T cell responses | baseline, Day 57
  percent of CD4 and CD8 T cells that produce IFNγ following exposure to overlapping peptide pool representing the vaccine-encoded receptor binding domain (RBD).
Effect of age on Geometric mean titer (GMT) in RA patients | baseline, Day 57
  Will be assessed by comparing RA treated with JAKs versus biologics versus RTX in age adjusted models.
Geometric mean titer (GMT) in RA versus age-matched controls | baseline, Day 57
  Will be assessed by comparing RA versus HC in age adjusted models.
Geometric mean titer (GMT) | baseline, Month 6 and Month 12
Percentage of patients who seroconverted | baseline, Day 57
  defined as a 4-fold increase in neutralizing antibody titer
Geometric mean fold rise (GMFR) of neutralizing antibody titer | baseline, Day 57
Effect of treatment on Geometric mean titer (GMT) in RA patients | baseline, Day 57
  Will be assessed by comparing RA treated with JAKs versus biologics versus RTX in age adjusted models.

CONTACTS AND LOCATIONS:
Overall Officials: Ines Colmegna, DR, Principal Investigator — RI-MUHC
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No